CLINICAL TRIAL: NCT06573216
Title: Clinical Trial on the Effectiveness and Safety of Blood Pressure Function System of Wrist Ambulatory Blood Pressure Monitor
Brief Title: Clinical Trial of Wrist Ambulatory Blood Pressure Monitor in Conformance With the EN ISO 81060-2:2018+AMD1:2020
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huawei Device Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-PPA0971CHN24011810332987
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood pressure measured by wrist ambulatory blood pressure monitor and mercury sphygmomanometer (Experimental)
  Interventions: Device: Wrist Ambulatory Blood Pressure Monitor

INTERVENTIONS:
Device: Wrist Ambulatory Blood Pressure Monitor — Comparing blood pressure measured by wrist blood pressure monitor with mercury sphygmomanometer .

SUMMARY:
The accuracy and safety of the Wrist Ambulatory Blood Pressure Recorder (Model: LCA-B10) were assessed according to the requirements of EN ISO 81060-2:2018 + AMD1:2020.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should voluntarily participate in the clinical trial and sign the informed consent form;
2. Subjects must be willing and able to follow the study procedures;
3. Subjects are over 18 years old whose wrist circumference should be within 13.0-21.0cm.

Exclusion Criteria:

1. Subjects with serious arrhythmias (atrial fibrillation, atrial flutter, ventricular flutter, ventricular fibrillation, ventricular tachycardia, borderline tachycardia, sinus arrest, pathological sinus syndrome, pacemaker rhythm) showed by electrocardiogram during screening period;
2. Subjects with sickle cell disease;
3. Subjects with prior mastectomy or arm lymph node dissection;
4. Subjects who are allergic to nylon, fluororubber or thermo-plastic polyurethane elastomer (TPU);
5. Subjects with wounds on the limb at the measurement site or inflammation of the wrist
6. Subjects who are undergoing intravenous fluid therapy, blood transfusion or other catheterization at the measurement site limb;
7. Subjects who have eaten, consumed alcohol, smoked cigarettes, or exercised vigorously 30 minutes prior to the trial;
8. Subjects who have participated in other clinical trials within 30 days that may affect this trial;
9. Subjects who, in the opinion of the investigator, should not participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure mean deviation and standard deviation- evaluation criterion 1 | 30 minutes
  The mean deviation and standard deviation between the blood pressure values measured by the investigational device and those obtained using the auscultatory method with the reference device. This calculation is performed on valid data pairsof subjects (n≥255).
  Evaluation criterion 1: The blood pressure mean deviation should not exceed ±5mmHg, and the standard deviation should not exceed 8mmHg.
Blood pressure mean deviation and standard deviation- evaluation criterion 2 | 30 minutes
  The mean deviation and standard deviation between the blood pressure values measured by the investigational device and those obtained using the auscultatory method with the reference device. This calculation is performed on the valid data group of all subjects (m≥85).
  Evaluation criterion 2: The blood pressure standard deviation within the valid data group (m ≥ 85) should not exceed the maximum allowable standard deviation corresponding to the mean deviation listed in Criterion 2 in section 5.2.4.1.2 b of ISO 81060-2:2018+AMD1:2020.
The mean deviation and standard deviation of blood pressure measurements under ambulatory blood pressure monitoring | 30 minutes
  The mean deviation and standard deviation of the blood pressure within the valid data group are calculated to evaluate whether the clinical accuracy of the investigational device meets the requirements outlined in ISO 81060-2:2018+AMD1:2020, specifically in section 5.2.4.1.2a).
  The blood pressure mean deviation should not exceed ±5mmHg, and the standard deviation should not exceed 8mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Bin Peng, Chenzhou, Hunan, China